CLINICAL TRIAL: NCT05779475
Title: An Observational Study of Patients With Moderate Parkinson's Disease
Acronym: TRANSCEND 1
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9001-4704; U1111-1254-1741 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Parkinson's disease: Participants will not receive any investigational treatment in this study. The participants will be treated with anti-Parkinson's disease medication according to local standard of care.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Participants will not receive any investigational treatment in this study.

SUMMARY:
The main purpose of this study is to follow and observe a group of people living with Parkinson's disease to see how study participation affects their signs and symptoms in the months after starting in the study. While taking part in this study participants will take their usual medication as prescribed. However, the study doctor may recommend adjustments to their medication to provide a better treatment of their Parkinson's disease. Participation will last from 3 up to 24 months. During visits to the clinic, the study doctor or study nurse will evaluate signs and symptoms of Parkinson's disease using several different assessments. At a minimum of 2 visits participants will be asked to undergo 'off'-assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 50-68 years (both inclusive) at the time of signing informed consent.
* Diagnosed with Parkinson's disease using the Movement Disorder Society (MDS) criteria (fulfilling the definition of clinically probable Parkinson's disease).
* Moderate Parkinson's disease, e.g. as defined by i) modified Hoehn and Yahr stage 2-3 in OFF state and ii) MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III total score greater than or equal to (≥) 30 in OFF state, both as judged by the investigator.
* Patient has symptoms that are not adequately controlled by existing oral anti-Parkinson's disease medications, i.e., having both ON and OFF periods, as judged by the investigator.
* Parkinson's disease duration greater than (>) 5 years and lesser than or equal to (≤) 12 years from diagnosis at the time of signing informed consent.
* Potential candidate for a future cell therapy transplantation, as judged by the investigator.
* Life expectancy >7 years as judged by the investigator.

Exclusion Criteria:

* Any atypical or secondary Parkinson's disease, or non-Parkinson's disease-suspected cause(s) of, or contributors to, parkinsonism, as judged by the investigator.
* Significant drug-induced dyskinesias as judged by the investigator, e.g., as defined by a score of > 2 in the Abnormal Involuntary Movement Scale (AIMS), in any body part in the ON state.
* Tremor-dominant Parkinson's disease, as judged by the investigator.
* Cognitive impairment predictive of dementia (including Parkinson's disease dementia) or other cognitive dysfunction as judged by the investigator, e.g., as defined by Montreal Cognitive Assessment (MoCA) score ≤ 24, or evidence of major neurocognitive disorder according to the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) criteria.
* Major medical or psychiatric disorder (e.g., depression (Montgomery-Asberg Depression Rating Scale (MADRS) >20) or psychosis), or other disease making the patient unsuited for participation in the study, as judged by the investigator.
* Treatment for dystonia or spasticity within 3 months of screening (Botox for a focal dystonia is allowed).
* Substantial neurological symptoms not accounted for by Parkinson's disease, including active seizure disorder, as judged by the investigator.

Ages: 50 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Parkinson's disease will be included. The participants will not receive any investigational treatment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2030-03-11 (Estimated); Study Completion 2030-03-11 (Estimated)

PRIMARY OUTCOMES:
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (motor score) in OFF state | From baseline (week 0) to end of study (13 to 104 weeks from baseline)
  Measured as score. MDS-UPDRS consists of 4 parts - has 65 items/questions in total. Part III assesses the motor function of the patient at the time of the visit conducted in both the OFF and ON state. Each item will receive a score ranging from 0 to 4, where 0 represents the absence of impairment and 4 represents the highest degree of impairment.

SECONDARY OUTCOMES:
Change in MDS-UPDRS Part III (motor score) in OFF state | From last medication adjustment (between week 0 and week 104) to end of study (13 to 104 weeks from baseline)
  Measured as score. MDS-UPDRS consists of 4 parts - has 65 items/questions in total. Part III assesses the motor function of the patient at the time of the visit conducted in both the OFF and ON state. Each item will receive a score ranging from 0 to 4, where 0 represents the absence of impairment and 4 represents the highest degree of impairment.
Is the patient interested in being considered for participation in a cell therapy transplantation study (yes/no) | At end of study (13 to 104 weeks from baseline)
  Measured as count of participants

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (8):
- United States (3):
  - Joe C.Wen & Fam CTR for Adv Care, Irvine, California
  - NYU Langone Health, New York, New York
  - NY Presbyt Hosp-W Cornell Med, New York, New York
- Keio University Hospital, Shinjuku-ku, Tokyo, Japan
- Sweden (2):
  - Neurologimottagningen Lund, Lund
  - Region Skane Skanes Universitetssjukhus, Lund
- United Kingdom (2):
  - Clinical Neuroscience, Cambridge
  - University of Cambridge - Clinical Neuroscience, Cambridge

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com